CLINICAL TRIAL: NCT05654181
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, 4-PERIOD, CROSSOVER, FIRST-IN-HUMAN STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF SINGLE ASCENDING ORAL DOSES OF PF-07328948 ADMINISTERED TO HEALTHY ADULT PARTICIPANTS
Brief Title: A First-in-human Study of Single Doses of PF-07328948 Which is Given to Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: C4921001
Record Dates: First submitted 2022-10-13; First posted 2022-12-16 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants will receive up to 4 dose levels of PF-07328948 single dose and up to 2 single doses of matching placebo. Doses will be administered as oral suspensions and each dose level is to be determined.
  Interventions: Drug: PF-07328948; Drug: Placebo
- Cohort 2 (Experimental): Participants will receive up to 4 dose levels of PF-07328948 single dose and up to 2 single doses of matching placebo. Doses will be administered as oral suspensions and each dose level is to be determined.
  Interventions: Drug: PF-07328948; Drug: Placebo
- Cohort 3 (Experimental): Participants will receive up to 4 dose levels of PF-07328948 single dose and up to 2 single doses of matching placebo. Doses will be administered as oral suspensions and each dose level is to be determined.
  Interventions: Drug: PF-07328948; Drug: Placebo

INTERVENTIONS:
Drug: PF-07328948 — investigational drug administered orally
Drug: Placebo — Placebo matching active drug administered orally

SUMMARY:
This study is the first clinical study with PF-07328948. The safety, tolerability, and plasma pharmacokinetics and pharmacodynamics of PF-07328948 after administration of escalating, single, oral doses will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants of non-childbearing potential and males must be 18 to 60 years of age, inclusive, at the time of signing the Informed Consent Document (ICD).
2. Female participants of non-childbearing potential and males who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

   * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
   * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBcAb, or HCVAb. Hepatitis B vaccination is allowed.
2. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
3. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
4. Receipt of a COVID-19 vaccine within 7 days before screening or within 7 days before any visit in which a safety lab is planned. Vaccination with a COVID 19 vaccine that occurs greater than 7 days from either screening or any visit in which a safety lab is planned is permitted.
5. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
6. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
7. Renal impairment as defined by an eGFR <75 mL/min/1.73m2 calculated using CKD EPI SCr formulas.
8. Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate age myocardial infarction, STT interval changes suggestive of myocardial ischemia, second- or third-degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the uncorrected QT interval is >450 ms, this interval should be rate corrected using the Fridericia method only and the resulting QTcF should be used for decision-making and reporting.
9. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * AST or ALT level ≥1.25× ULN;
   * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ULN.
10. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
11. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4921001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 20 participants were enrolled, and received at least one dose of study intervention.
Groups:
- PF-07328948 10 mg, PF-07328948 30 mg, PF-07328948 100 mg, Placebo; PF-07328948 10 mg, PF-07328948 30 mg, Placebo, PF-07328948 300 mg; PF-07328948 10 mg, Placebo, PF-07328948 100 mg, PF-07328948 300 mg; Placebo, PF-07328948 30 mg, PF-07328948 100 mg, PF-07328948 300 mg: Participants were assigned to Cohort 1 in four sequences (Sequence: PF-07328948 10 mg, 30 mg, 100 mg, placebo; Sequence: 10 mg, 30 mg, placebo, 300 mg; Sequence: 10 mg, placebo, 100 mg, 300 mg; and Sequence: placebo, 30 mg, 100 mg, 300 mg).
- PF-07328948 750 mg, PF-07328948 F mg, PF-07328948 G mg, Placebo; Placebo, PF-07328948 F mg, PF-07328948 G mg, PF-07328948 H mg: Participants assigned to sentinel dose in Cohort 2 Period 1 were terminated after Period 1. (The letters 'F', 'G' and 'H' stand for the planned escalating doses.)
- PF-07328948 300 mg, PF-07328948 750 mg, PF-07328948 1500 mg, PF-07328948 750 mg (Fed); PF-07328948 300 mg, PF-07328948 750 mg, Placebo, PF-07328948 750 mg (Fed); PF-07328948 300 mg, Placebo, PF-07328948 1500 mg, Placebo (Fed); Placebo, PF-07328948 750 mg, PF-07328948 1500 mg, PF-07328948 750 mg (Fed): Participants were assigned to Cohort 3 in four sequences (Sequence: 300 mg, 750 mg, 1500 mg, 750 mg [fed]; Sequence: 300 mg, 750 mg, placebo, 750 mg [fed]; Sequence: 300 mg, placebo, 1500 mg, placebo [fed]; and Sequence: placebo, 750 mg, 1500 mg, 750 mg [fed]).
Period: Overall Study
Arm/Group | PF-07328948 10 mg, PF-07328948 30 mg, PF-07328948 100 mg, Placebo | PF-07328948 10 mg, PF-07328948 30 mg, Placebo, PF-07328948 300 mg | PF-07328948 10 mg, Placebo, PF-07328948 100 mg, PF-07328948 300 mg | Placebo, PF-07328948 30 mg, PF-07328948 100 mg, PF-07328948 300 mg | PF-07328948 750 mg, PF-07328948 F mg, PF-07328948 G mg, Placebo | Placebo, PF-07328948 F mg, PF-07328948 G mg, PF-07328948 H mg | PF-07328948 300 mg, PF-07328948 750 mg, PF-07328948 1500 mg, PF-07328948 750 mg (Fed) | PF-07328948 300 mg, PF-07328948 750 mg, Placebo, PF-07328948 750 mg (Fed) | PF-07328948 300 mg, Placebo, PF-07328948 1500 mg, Placebo (Fed) | Placebo, PF-07328948 750 mg, PF-07328948 1500 mg, PF-07328948 750 mg (Fed)
Started | 3 | 2 | 2 | 2 | 1 | 1 | 2 | 3 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 2 | 1 | 2 | 2
Not Completed | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-07328948 10 mg, PF-07328948 30 mg, PF-07328948 100 mg, Placebo | PF-07328948 10 mg, PF-07328948 30 mg, Placebo, PF-07328948 300 mg | PF-07328948 10 mg, Placebo, PF-07328948 100 mg, PF-07328948 300 mg | Placebo, PF-07328948 30 mg, PF-07328948 100 mg, PF-07328948 300 mg | PF-07328948 750 mg, PF-07328948 F mg, PF-07328948 G mg, Placebo | Placebo, PF-07328948 F mg, PF-07328948 G mg, PF-07328948 H mg | PF-07328948 300 mg, PF-07328948 750 mg, PF-07328948 1500 mg, PF-07328948 750 mg (Fed) | PF-07328948 300 mg, PF-07328948 750 mg, Placebo, PF-07328948 750 mg (Fed) | PF-07328948 300 mg, Placebo, PF-07328948 1500 mg, Placebo (Fed) | Placebo, PF-07328948 750 mg, PF-07328948 1500 mg, PF-07328948 750 mg (Fed) | Total
Number analyzed (Participants) | 3 | 2 | 2 | 2 | 1 | 1 | 2 | 3 | 2 | 2 | 20
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 1 | 2 | 2 | 2 | 1 | 1 | 1 | 3 | 0 | 0 | 13
  45-60 years | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Male | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 3 | 2 | 0 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 3 | 1 | 1 | 2 | 1 | 1 | 1 | 3 | 1 | 2 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5
  Black or African American | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 2 | 0 | 1 | 9
  Asian | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Multiple | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Not reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An adverse event is considered a TEAE if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the end of the study were flagged as TEAEs. The algorithm did not consider any events that started prior to the first dose date. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Day 1-8 per period, along with the 28-35 day post-final dose follow-up
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants assigned to Cohort 1, Cohort 2, and Cohort 3 received placebo.
- Placebo (Fed): Participants assigned to Cohort 3 received placebo (fed).
- PF-07328948 10 mg: Participants assigned to Cohort 1 received PF-07328948 10 mg.
- PF-07328948 30 mg: Participants assigned to Cohort 1 received PF-07328948 30 mg.
- PF-07328948 100 mg: Participants assigned to Cohort 1 received PF-07328948 100 mg.
- PF-07328948 300 mg: Participants assigned to Cohort 1 and Cohort 3 received PF-07328948 300 mg.
- PF-07328948 750 mg: Participants assigned to Cohort 2 and Cohort 3 received PF-07328948 750 mg.
- PF-07328948 750 mg (Fed): Participants assigned to Cohort 3 received PF-07328948 750 mg (fed).
- PF-07328948 1500 mg: Participants assigned to Cohort 3 received PF-07328948 1500 mg.
Arm/Group | Placebo | Placebo (Fed) | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
Number analyzed (Participants) | 13 | 2 | 6 | 5 | 5 | 12 | 7 | 5 | 6
Participants
  All-causality AEs | 3 | 1 | 3 | 2 | 1 | 5 | 3 | 1 | 2
  Treatment-related AEs | 1 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 1
  All-causality SAEs | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related SAEs | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Meeting Pre-Defined Categorical Criteria Without Regard to Baseline Abnormality
Description: Pre-defined categorical criteria for laboratory abnormalities included: lymphocytes/Leukocytes <0.8 x lower limit of normal (LLN) or >1.2 x upper limit of normal (ULN); Neutrophils <0.8 x LLN; Neutrophils/Leukocytes <0.8 x LLN; Eosinophils/Leukocytes >1.2 x ULN; Monocytes/Leukocytes >1.2 x ULN; Bilirubin >1.5 x ULN; Indirect Bilirubin >1.5 x ULN; Ketones (Scalar) ≥1; URINE Hemoglobin (Scalar) ≥1; URINE Bilirubin (Scalar) ≥1; Leukocyte Esterase (Scalar) ≥1; and Bacteria (/HPF) >20.
Time Frame: Day 1-8 per period, along with the 28-35 day post-final dose follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Placebo (Fed) | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
Number analyzed (Participants) | 13 | 2 | 6 | 5 | 5 | 12 | 7 | 5 | 6
Participants | 0 | 0 | 1 | 2 | 1 | 3 | 3 | 1 | 2

3. Primary Outcome: Number of Participants With Vital Signs Abnormalities Meeting Pre-Defined Categorical Criteria
Description: Vital signs categorical criteria: 1) supine systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); 2) supine diastolic blood pressure (DBP) <50 mmHg; 3) supine pulse rate <40 or >120 beats per minute (bpm); 4) change from baseline (increase or decrease) in supine SBP greater than or equal to (≥) 30 mmHg; 5) change from baseline (increase or decrease) in supine DBP ≥ 20 mmHg.
Time Frame: Day 1-8 per period, along with the 28-35 day post-final dose follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Placebo (Fed) | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
Number analyzed (Participants) | 13 | 2 | 6 | 5 | 5 | 12 | 7 | 5 | 6
Participants
  SBP <90 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Change from baseline in SBP ≥30 mmHg decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change from baseline in SBP ≥30 mmHg increase | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  DBP <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change from baseline in DBP ≥20 decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change from baseline in DBP ≥20 increase | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Pulse rate < 40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate > 120 bpm | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Meeting Pre-Defined Categorical Criteria
Description: ECG categorical criteria: 1. PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): a) ≥300 millisecond (msec), b) ≥25% increase when baseline is > 200 msec or ≥50% increase when baseline is less than or equal to (≤) 200 msec.
  2. QRS interval (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): a) ≥140 msec, b) ≥50% increase from baseline.
  3. QTcF interval (QT corrected using the Fridericia formula): a) >450 msec and ≤480 msec, b) >480 msec and ≤500 msec, c) >500 msec, d) >30 msec and ≤60 msec increase from baseline, e) >60 msec increase from baseline
Time Frame: Day 1-8 per period, along with the 28-35 day post-final dose follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Placebo (Fed) | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
Number analyzed (Participants) | 13 | 2 | 6 | 5 | 5 | 12 | 7 | 5 | 6
Participants
  PR interval ≥300 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  %Change in PR interval ≥25/50% increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS interval ≥140 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  %Change in QRS interval ≥50% increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval >450 and ≤480 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval >480 and ≤500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval >500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change in QTcF interval >30 and ≤60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change in QTcF interval >60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters (ECG Mean Heart Rate)
Description: Maximum increase from baseline in ECG Mean Heart Rate was reported.
Time Frame: Day 1-8 per period, along with the 28-35 day post-final dose follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | Placebo (Fed) | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
Number analyzed (Participants) | 13 | 2 | 6 | 5 | 5 | 12 | 7 | 5 | 6
bpm | 9.52 (5.179) | 12.45 (2.616) | 9.75 (2.752) | 12.88 (3.321) | 8.36 (4.821) | 16.32 (14.132) | 15.53 (3.892) | 16.32 (4.437) | 13.42 (3.845)

6. Secondary Outcome: Maximum Concentration Observed in Plasma (Cmax)
Description: Maximum observed plasma PF-07328948 concentration. Observed directly from data.
Time Frame: Pre-dose (0 hours) and 0.5 hours, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 8 hours and 12 hours post Day 1 dosing of each Period (Periods 1-4)
Population: All participants randomly assigned to study intervention and who received at least 1 dose of study intervention and had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
Number analyzed (Participants) | 6 | 5 | 5 | 12 | 7 | 5 | 6
nanogram per milliliter (ng/mL) | 294.7 (111) | 1549 (11) | 7049 (18) | 19100 (25) | 40220 (33) | 37440 (13) | 61030 (44)

7. Secondary Outcome: Time to Achieve Cmax (Tmax)
Description: Observed directly from data as time of first occurrence.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
Number analyzed (Participants) | 6 | 5 | 5 | 12 | 7 | 5 | 6
hours (hr) | 1.10 [1.00 to 3.00] | 3.00 [1.00 to 4.00] | 2.00 [1.50 to 3.00] | 3.00 [1.50 to 4.00] | 3.02 [3.00 to 4.02] | 4.00 [2.00 to 4.03] | 3.04 [2.00 to 8.03]

8. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Measured Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration. It was determined by using linear/Log trapezoidal method.
Time Frame: as for outcome 6
Population: All participants randomly assigned to study intervention and who received at least 1 dose of study intervention and had at least 1 of the PK parameters of interest calculated. Number of participants analyzed = participants who were evaluable for this OM and contributed to the summary statistics of this OM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
Number analyzed (Participants) | 3 | 5 | 5 | 12 | 7 | 5 | 6
nanogram*hour per milliliter (ng*hr/mL) | 0.0000 (NA) — The CV is NA (not reportable) for the PF-07328948 10 mg as all 3 individuals had values of 0 with mean of 0 and CV is undefinable. | 4396 (11) | 35030 (23) | 110200 (30) | 363600 (24) | 409300 (26) | 742700 (24)

9. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUCinf)
Description: Area under the plasma concentration-time curve from time 0 extrapolated to infinite time. AUCinf = AUClast + (Clast*/kel), where Clast* is the predicted plasma concentration at the last quantifiable timepoint estimated from the log-linear regression analysis, and Kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve, AUClast = Area under the plasma concentration time-curve from zero to the last measured concentration.
Time Frame: as for outcome 6
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
Number analyzed (Participants) | 0 | 0 | 4 | 11 | 7 | 5 | 4
nanogram*hour per milliliter (ng*hr/mL) |  |  | 39050 (19) | 114300 (32) | 378000 (26) | 427600 (29) | 774600 (28)

10. Secondary Outcome: Terminal Half-Life (t1/2) of PF-07328948
Description: Terminal elimination half-life. t1/2 = Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log linear decline will be used in the regression.
Time Frame: as for outcome 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
Number analyzed (Participants) | 0 | 0 | 4 | 11 | 7 | 5 | 4
hours (hr) |  |  | 11.58 (4.2565) | 9.941 (2.4980) | 16.13 (6.5277) | 16.90 (5.1749) | 15.90 (5.5106)

11. Primary Outcome: Change From Baseline in ECG Parameters (PR Interval, QRS Duration, and QTcF Interval)
Description: Maximum increase from baseline in PR Interval, QRS Duration, and QTcF Interval was reported.
Time Frame: Day 1-8 per period, along with the 28-35 day post-final dose follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | Placebo (Fed) | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
Number analyzed (Participants) | 13 | 2 | 6 | 5 | 5 | 12 | 7 | 5 | 6
msec
  Maximum increase from baseline in PR Interval (msec) | 5.15 (5.536) | 5.10 (1.414) | 2.30 (4.260) | 2.12 (2.139) | 0.80 (4.540) | 3.93 (3.215) | 6.86 (8.703) | 10.00 (5.477) | 5.73 (1.952)
  Maximum increase from baseline in QRS Duration (msec) | 3.54 (3.227) | 10.60 (3.111) | 1.73 (2.534) | 2.44 (2.014) | 0.14 (0.969) | 4.11 (2.858) | 0.91 (3.065) | 6.20 (3.251) | 4.40 (5.303)
  Maximum increase from baseline in QTcF Interval (msec) | 6.95 (5.949) | 7.40 (3.960) | 3.10 (4.900) | 3.40 (2.879) | 1.78 (6.634) | 2.84 (4.702) | 6.90 (11.844) | 1.50 (5.236) | 8.47 (8.281)

ADVERSE EVENTS:
Time Frame: Day 1-8 per period, along with the 28-35 day post-final dose follow-up
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | Placebo (Fed) | PF-07328948 10 mg | PF-07328948 30 mg | PF-07328948 100 mg | PF-07328948 300 mg | PF-07328948 750 mg | PF-07328948 750 mg (Fed) | PF-07328948 1500 mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/2 | 0/6 | 0/5 | 0/5 | 0/12 | 0/7 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/2 | 0/6 | 0/5 | 0/5 | 0/12 | 0/7 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 3/13 | 1/2 | 3/6 | 2/5 | 1/5 | 5/12 | 3/7 | 1/5 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Placebo (Fed) (N=2) | PF-07328948 10 mg (N=6) | PF-07328948 30 mg (N=5) | PF-07328948 100 mg (N=5) | PF-07328948 300 mg (N=12) | PF-07328948 750 mg (N=7) | PF-07328948 750 mg (Fed) (N=5) | PF-07328948 1500 mg (N=6)
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Placebo (Fed) (N=2) | PF-07328948 10 mg (N=6) | PF-07328948 30 mg (N=5) | PF-07328948 100 mg (N=5) | PF-07328948 300 mg (N=12) | PF-07328948 750 mg (N=7) | PF-07328948 750 mg (Fed) (N=5) | PF-07328948 1500 mg (N=6)
Application site dermatitis (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT05654181/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT05654181/SAP_001.pdf